CLINICAL TRIAL: NCT00979433
Title: Bubble CPAP vs. Conventional CPAP Following Extubation in Preterm Very Low Birth Weight (VLBW) Infants: A Randomized Controlled Trial
Brief Title: Bubble Continuous Positive Airway Pressure (CPAP) With Conventional CPAP for Extubation in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ramesh K Agarwal, Associate Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-74
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Extubation Failure
Keywords: Extubation failure; Continuous positive airway pressure; Bubble CPAP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bubble CPAP (Experimental): All neonates randomised to bubble CPAP will be put on Bubble CPAP following initial extubation in first week of life.
  Interventions: Device: Bubble CPAP
- Conventional CPAP (Other): All neonates randomly allocated to conventional/ventilator derived CPAP.
  Interventions: Device: Conventional CPAP

INTERVENTIONS:
Device: Bubble CPAP — Bubble CPAP will be delivered using Fischer & Paykel CPAP system with a starting flow of 6 liters/minute. CPAP will be initially started at a pressure of 5 - 6 cm H2O and fraction of inspired oxygen (FiO2) of 0.4 - 0.5. which will be adjusted to maintain oxygen saturation (SpO2) between 87 and 93%.
  Other Names: Fisher & Paykel Bubble CPAP System
  Arms: Bubble CPAP
Device: Conventional CPAP — Conventional CPAP will be delivered using Argyle CPAP (Sherwood Medical Company, Mexico) short nasal prongs with warm, humidified gas used (34-37°C) through a thermo-statically controlled humidifier, flow @ 4-8 L/min from either SLE 2000 pressure-controlled continuous flow ventilator (Specialized Laboratory Equipment, UK) or Baby log 8000 volume guarantee ventilator.
  Arms: Conventional CPAP

SUMMARY:
The objective of this study is to evaluate whether CPAP delivered by bubble CPAP resulted in a greater proportion of infants being successfully extubated when compared with management with ventilator derived CPAP.

DETAILED DESCRIPTION:
There have been no published randomized trials comparing extubation failure rates of Bubble CPAP with conventional ventilator derived CPAP. Infants of gestation <32 weeks and of birth weight less than 1500 grams considered by the treating team to be ready for the initial extubation within first week of life were screened for enrolment. All eligible neonates were randomly allocated to bubble CPAP or conventional CPAP.The purpose of this study is to compare whether infants on Bubble CPAP had more chances of successful extubation as compared to infants put on Conventional CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Gestation less than 32 weeks
* Birth weight less than 1500 g
* Age less than seven days
* First extubation attempt.

Exclusion Criteria:

* A neonate having any of the following will be excluded from the study-
* Severe birth asphyxia defined as need for chest compression for more than 30 seconds
* Suspected congenital neuromuscular disorder
* Major congenital malformation
* Grade 3/4 interventricular haemorrhage
* Hydrops.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Extubation failure - defined as need for reintubation and mechanical ventilation for any reason within 72 hours of initial extubation | Till 72 hours after extubation

SECONDARY OUTCOMES:
Time to extubation failure in hours. | till extubation failure within first 72 hours after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Vinod K Paul, MD PhD, Study Chair — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Sucheta Yadav, MBBS, Principal Investigator — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Mari J Sankar, MD, DM, Study Chair — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Ramesh Agarwal, MD, DM, Study Chair — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India